CLINICAL TRIAL: NCT04047771
Title: A Phase I Study Evaluating the Safety, Tolerability and Pharmacokinetics of SCB-313, Recombinant Human Tumor Necrosis Factor-Related Apoptosis-Inducing Ligand-Trimer Fusion Protein, for the Treatment of Subjects With Peritoneal Carcinomatosis
Brief Title: A Phase I Study Evaluating SCB-313 for the Treatment of Subjects With Peritoneal Carcinomatosis
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: terminated
Sponsor: Sichuan Clover Biopharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CLO-SCB-313-CHN-003
Record Dates: First submitted 2019-08-05; First posted 2019-08-07 (Actual); Last update posted 2023-04-12 (Actual); Status verified 2023-04

CONDITIONS: Peritoneal Carcinomatosis
MeSH Terms: conditions — Peritoneal Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SCB-313 (Experimental)
  Interventions: Drug: SCB-313

INTERVENTIONS:
Drug: SCB-313 — Intraperitoneal injection, 3 doses on D1,D4,D7，21 days for 1 cycle
  Other Names: recombinant human TRAIL-Trimer fusion protein

SUMMARY:
To evaluate the safety and tolerability of SCB-313 in patients with peritoneal carcinomatosisa, to determine the maximum tolerated dose (MTD) and/or extended study recommended dose (RDE) for SCB-313 intraperitoneal injection, providing a basis for dosing regimen and dose choosing in clinical trial subsequently.

ELIGIBILITY:
Inclusion Criteria:

1. Be able to understand and voluntarily sign written informed consent.
2. Male or female subjects, age ≥18, ≤75 years.
3. Confirmed by histopathology or cytopathology, any primary or secondary malignant peritoneal carcinomatosis subject.
4. Progression after standard treatment, or inability to tolerate standard treatment, or no standard treatment.
5. ECOG status 0 to 2 or KPS status > 60
6. CT-PCI (Peritoneal Carcinomatosis Index) status ≥ 15
7. Life expectancy of at least 3 months.
8. No serious hematologic, hepatic, renal dysfunction, comply with the following laboratory test results:

   1. Hematology: white blood cell count >3*109/L, absolute neutrophil count ≥1.5*109/L, platelets > 75*109/L, hemoglobin > 90 g/L.
   2. Liver function: aspartate aminotransferase and alanine aminotransferase ≤ 3 times ULN, Alkaline phosphatase (ALP) ≤ 2.5 times ULN; serum total bilirubin (TBIL) ≤ 1.5 times ULN.
   3. Renal function: Creatinine clearance calculated according to the Cockcroft-Gault formula ≥ 50 mL/min.
9. All adverse events from previous system anticancer treatment return to baseline or ≤ grade 1 (except for alopecia and vitiligo, neuropathy which induced by previous anticancer therapy status stable or ≤ grade 2).
10. Male or female subjects undergo effective contraception during treatment and within 6 months after last dose.

Exclusion Criteria:

1. Previous treatment with TRAIL pathway drug.
2. Malignant cancer diseases other than malignant peritoneal carcinomatosis in this study (Exceptions include: a cured malignant cancer without relapse within 3 years prior to the study enrollment, completely resected basal cells and squamous cell skin cancer, and any type of carcinoma in situ).
3. Primary lesion invades the central nervous system (CNS) with symptoms develop, status unstable or require high dose steroids (e.g. dexamethasone ≥ 10 mg or equivalent dose) to control.
4. Abnormal HBV examination, anti-HCV positive, anti-HIV antibody positive or other serious infections requiring systemic treatment within 4 weeks prior to first dosing (e.g. virus, bacteria or fungus).
5. Use the following concomitant therapy before dosing:

   1. Use drug that prolongs the QT interval and/or associated with the risk of torsades de pointes ventricular tachycardia (TdP) within 7 days prior to first dosing.
   2. Use amiodarone within 90 days prior to first dosing.
6. Impaired heart function or clinically significant cardiovascular disease, including any of the following:

   1. Cerebrovascular accident/stroke (within 6 months prior to enrollment).
   2. Myocardial infarction (within 6 months prior to enrollment).
   3. Unstable angina, congestive heart failure (New York Heart Association grade ≥ II) or severe arrhythmia requiring medication (including QT/QTc interval extension >480 msec, installation of pacemakers, etc.).
   4. Left ventricular ejection fraction < 50% as determined by echocardiography.
7. Active bleeding history or gastrointestinal perforation risk within 4 weeks before enrollment, or not healed from recent surgery.
8. Received anticancer treatment within following specified time before first dosing:

   1. Received medical treatment ≤ 4 weeks or 5 times known drug half-life (whichever is longer).
   2. Underwent major surgery within ≤ 4 weeks before first dosing.
9. Residual adverse events from previous treatment≥ grade 2.
10. Known to have alcohol and/or drug dependence.
11. Previous clear history of neurological or mental disorders, such as epilepsy, poor compliance
12. Female subjects with positive blood pregnancy tests or during lactation.
13. Previously allergic to macromolecular protein drugs or proteins or Quincke's edema (Kunke edema, also known as angioedema) or allergic to any component of the SCB 313.
14. Known history of infection with human immunodeficiency virus, or other acquired, innate immune deficiency diseases, or history of organ transplantation.
15. Vaccination within ≤ 4 weeks prior to first dosing, or planning live vaccination.
16. For other reasons according to investigators, not suitable for participation in the trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2019-09-10 (Actual); Primary Completion 2022-05-05 (Actual); Study Completion 2022-05-05 (Actual)

PRIMARY OUTCOMES:
Dose Limiting Toxicity (DLT) | 21 days after first dosing
  DLT
Occurrence of adverse events (AEs) and serious adverse events (SAEs) | 21 days after first dosing
  AEs

SECONDARY OUTCOMES:
Immunogenicity | 28 days after last dosing
  Occurrence of binding and neutralizing anti-SCB-313 antibodies
Pharmacokinetics (Cmax) | Up to 24 hours after dosing
  Maximum SCB-313 concentration
Pharmacokinetics (tmax) | Up to 24 hours after dosing
  Time to Cmax of SCB-313
Pharmacokinetics ([AUC]0-24) | Up to 24 hours after dosing
  Area under SCB-313 concentration time curve from zero to 24 hours
Pharmacokinetics (AUC 0-inf) | Up to 24 hours after dosing
  Area under curve from time 0 extrapolated to infinity

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Shijitan Hospital Capital Medical University, Beijing, Beijing Municipality, China